CLINICAL TRIAL: NCT06096597
Title: Amniotic Membrane Therapy for Interstitial Cystitis/Painful Bladder Syndrome (IC/PBS): a Prospective, Double-Blind, Randomized Controlled Trial
Brief Title: Amniotic Membrane Therapy for Interstitial Cystitis/Painful Bladder Syndrome
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: David Sheyn (Other)
Responsible Party: Sponsor-Investigator, David Sheyn, Physician, UH Hospitals, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY20231301; NCT06104787 (obsolete NCT alias)
Record Dates: First submitted 2023-10-17; First posted 2023-10-24 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Interstitial Cystitis; Painful Bladder Syndrome; Painful Bladder Syndrome (PBS)
Keywords: interstitial cystitis; painful bladder syndrome
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: At time of surgery, the surgeon will be given a sealed envelope containing a sterile syringe of either 10 mL of 0.9% preservative-free sodium chloride or 100 mg of commercially available micronized AM (Clarix Flo; BioTissue, Miami, FL) diluted in 10 mL of 0.9% preservative-free sodium chloride
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amniotic Membrane Therapy (Experimental): Under general anesthesia, cystoscopy will be performed. A needle will be inserted into the detrusor muscle to a depth of approximately 2 mm. 100mg of commercially available micronized amniotic membrane (Clarix Flo; BioTissue, Miami, FL) diluted in 10 mL of 0.9% preservative-free sodium chloride, and 0.5 mL of the solution will be injected into 20 equally spaced sites into the posterior and lateral walls of the bladder, sparing the dome and the trigone.
  Interventions: Drug: Clarix Flo
- Placebo (Placebo Comparator): Under general anesthesia, cystoscopy will be performed. A needle will be inserted into the detrusor muscle to a depth of approximately 2 mm. 0.5 mL of 10 mL of 0.9% preservative-free sodium chloride will be injected into 20 equally spaced sites into the posterior and lateral walls of the bladder, sparing the dome and the trigone.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clarix Flo — 100 mg of commercially available micronized amniotic membrane (Clarix Flo; BioTissue, Miami, FL) diluted in 10 mL of 0.9% preservative-free sodium chloride
  Arms: Amniotic Membrane Therapy
Drug: Placebo — 10 mL of 0.9% preservative-free sodium chloride
  Arms: Placebo

SUMMARY:
Interstitial cystitis/painful bladder syndrome (IC/PBS) is a clinical syndrome in which patients report symptoms of bladder and/or pelvic pain with pressure and/ or discomfort associated with urinary frequency and urgency.

The primary objective of this study is to determine the efficacy of amniotic membrane therapy in patients with interstitial cystitis/painful bladder syndrome (IC/PBS) as defined by clinically-significant improvement in validated symptom questionnaires.

DETAILED DESCRIPTION:
Interstitial cystitis/painful bladder syndrome (IC/PBS) is a clinical syndrome in which patients report symptoms of bladder and/or pelvic pain with pressure and/or discomfort associated with urinary frequency and urgency. These symptoms vary in severity and are known to cause significant impact on quality of life. Current recommended therapies include behavior modifications, stress management practices, physical therapy, oral pharmacologic pain management agents, intravesical instillations, hydrodistension, fulguration of bladder lesions and/or triamcinolone injections, intradetrusor onabotulinumtoxin A injections, neuromodulation, and major surgery.

Amniotic membranes, Clarix FLO™, have been used to assist in wound healing in many fields of medicine, and its use has evolved over the last century to various applications in regenerative medicine. A novel study using amniotic membranes for bladder therapy has showing promising preliminary results in a small cohort study of 10 females with recalcitrant IC/PBS. These women underwent intradetrusor injections of micronized amniotic membranes and had significant improvement of voiding symptoms and bladder pain over 3 months with no adverse events. No randomized controlled trials (RCT) of amniotic bladder therapy have been conducted to date. The proposed study would be the first RCT assessing the efficacy of amniotic membrane injections with Clarix FLO™ and has the potential to make significant impacts in the management and treatment of patients with IC/PBS.

Clarix FLO™ is a sterile, particulate human amniotic membrane and umbilical cord tissue product that is aseptically processed in compliance with current Good Tissue Practices from the same donated human tissue (placenta) after determination of eligibility and placenta/cord suitability. Amniotic Membrane and Umbilical Cord products are currently designated by the FDA as tissue products under PHS Act 361 HCT/P (human cells, tissues and cellular and tissue-based products). Clarix FLO™ does not contain living cells.

Patients will then be followed with clinical evaluation and questionnaires repeated at 2, 4, 8 and 12 weeks post-operatively. Additional urine culture and post void residuals will be repeated at 2 and 4 weeks post-operatively. Primary Objective: Determine the efficacy of amniotic bladder therapy (ABT) in patients with interstitial cystitis/painful bladder syndrome (IC/PBS) as defined by clinically-significant improvement

- Clinically-meaningful indicator defined as: 5 point reduction in Interstitial Cystitis Symptom Index (ICSI)

Secondary Objectives:

* Characterize duration of effect of ABT using clinical evaluation and the following questionnaires:
* Interstitial Cystitis Symptom Index (ICSI)
* Interstitial Cystitis Problem Index (ICPI)
* Bladder Pain/Interstitial Cystitis Symptom Score (BPIC-SS)
* Overactive Bladder Assessment Tool
* PUF
* SF-12 Health Survey
* Determine if there are any adverse effects of ABT, such as urinary tract infections or acute urinary retention.

Hypothesis: ABT in patients with PBS improves clinical outcomes

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Female
* English Speaking
* Diagnosis of IC/PBS
* Have failed at least one prior treatment for IC/PBS

Exclusion Criteria:

* Patients less than 18 years of age
* Unable to provide consent
* Non-English speaking
* Patients with known anatomical malformations of the ureters, bladder, or urethra

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Interstitial Cystitis Symptom Index (ICSI) score | To be completed pre-operatively and at 2, 4, 8 and 12 weeks post-operatively
  Evaluate for clinically-meaningful reduction in symptoms as defined as a 5 point reduction in Interstitial Cystitis Symptom Index (ICSI)

SECONDARY OUTCOMES:
Change in Interstitial Cystitis Symptom Index Questionnaire | To be completed pre-operatively and at 2, 4, 8 and 12 weeks post-operatively
  To determine the change in interstitial cystitis symptoms in participants who received amniotic membrane injection versus placebo injection (saline) as measured using the Interstitial Cystitis Symptom Index (ICSI).
Change in Interstitial Cystitis Problem Index Questionnaire | To be completed pre-operatively and at 2, 4, 8 and 12 weeks post-operatively
  To determine the change in interstitial cystitis symptoms in participants who received amniotic membrane injection versus placebo injection (saline) as measured using the Interstitial Cystitis Problem Index (ICPI).
Change in Bladder Pain/ Interstitial Cystitis Symptom Score | To be completed pre-operatively and at 2, 4, 8 and 12 weeks post-operatively
  To determine the change in interstitial cystitis symptoms in participants who received amniotic membrane injection versus placebo injection (saline) as measured using the Bladder Pain/Interstitial Cystitis Symptom Score (BPIC-SS).
Change in Overactive Bladder Assessment Tool Scores | To be completed pre-operatively and at 2, 4, 8 and 12 weeks post-operatively
  To determine the change in interstitial cystitis symptoms in participants who received amniotic membrane injection versus placebo injection (saline) as measured using the Overactive Bladder Assessment Tool
Change in SF-12 Health Survey Scores | To be completed pre-operatively and at 2, 4, 8 and 12 weeks post-operatively
  To determine the change in interstitial cystitis symptoms in participants who received amniotic membrane injection versus placebo injection (saline) as measured using the SF-12 Health Survey
Change in Pelvic Pain and Urgency/ Frequency (PUF) Patient Symptom Scale (PUF) Scores | To be completed pre-operatively and at 2, 4, 8 and 12 weeks post-operatively
  To determine the change in interstitial cystitis symptoms in participants who received amniotic membrane injection versus placebo injection (saline) as measured using the PUF Questionnaire
Change in number of urinary tract infections as measured by medical record review | To be completed pre-operatively and at 2, 4, 8 and 12 weeks post-operatively
  As defined by symptoms of urinary tract infection and positive urine culture

CONTACTS AND LOCATIONS:
Overall Officials: David Sheyn, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals, Clevleand, Ohio, United States

IPD SHARING:
Plan to Share IPD: No